CLINICAL TRIAL: NCT02202902
Title: Evaluation of Cardiac Steatosis in Cushing's Syndrome. A 1H-Magnetic Resonance Spectroscopy Study
Brief Title: Cardiac Steatosis in Cushing's Syndrome
Acronym: CORTICOEUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AOR12017; 2013-A01023-42 (Other: IDRCB)
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Endocrine System Disease; Cardiovascular Imaging
Keywords: Cushing's syndrome; cardiac steatosis; intramyocardial triglyceride content; 1H magnetic resonance spectroscopy and cardiac magnetic resonance imaging; Left Ventricularly hypertrophy
MeSH Terms: conditions — Endocrine System Diseases; Cushing Syndrome | interventions — Lead; Aftercare; Detection Algorithms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 : 1H magnetic resonance spectroscopy and CMRI (Experimental): Group 1 : Cushing's syndrome patients with diabetes mellitus or glucose intolerance
  Interventions: Other: 1H magnetic resonance spectroscopy and CMRI
- Group 2 : 1H magnetic resonance spectroscopy and CMRI (Experimental): Group 2: Cushing's syndrome patients with normal glucose intolerance
  Interventions: Other: 1H magnetic resonance spectroscopy and CMRI
- Group 3 : 1H magnetic resonance spectroscopy and CMRI (Experimental): age-, sex- and BMI-matched healthy volunteers
  Interventions: Other: 1H magnetic resonance spectroscopy and CMRI

INTERVENTIONS:
Other: 1H magnetic resonance spectroscopy and CMRI — Metabolic status of the patients evaluated by an OGTT (measuring plasma glucose, insulin and plasma nonesterified fatty acids concentrations) and myocardial Imaging and spectroscopy will be performed before and 6 month after treatment
  Other Names: Before and after Treatment
  Arms: Group 1 : 1H magnetic resonance spectroscopy and CMRI; Group 2 : 1H magnetic resonance spectroscopy and CMRI
Other: 1H magnetic resonance spectroscopy and CMRI — Metabolic status of the patients evaluated by an OGTT (measuring plasma glucose, insulin and plasma nonesterified fatty acids concentrations) and myocardial Imaging and spectroscopy will be performed before treatment
  Other Names: Once
  Arms: Group 3 : 1H magnetic resonance spectroscopy and CMRI

SUMMARY:
This study aims at evaluating the myocardial triglyceride content and cardiac structure and function, using 1H magnetic resonance spectroscopy and cardiac magnetic resonance imaging, in patients with Cushing's syndrome before and after treatment and in age-, sex- and BMI-matched healthy volunteers. The investigators make the hypothesis that Cushing's syndrome patients compared to healthy subjects present with excess lipid storage in cardiac myocytes, reversible upon correction of hypercortisolism.

DETAILED DESCRIPTION:
Despite skeletal muscle atrophy, Cushing's syndrome patients have an increased Left Ventricular mass, reversible upon correction of the hypercortisolism. This may be due to cardiac steatosis, previously demonstrated in patients with diabetes mellitus. This study aims at evaluating the myocardial triglyceride content and cardiac structure and function, using 1H magnetic resonance spectroscopy and cardiac magnetic resonance imaging (CMRI), in patients with Cushing's syndrome and in age-, sex- and BMI-matched healthy volunteers. The patients will be stratified into two groups in function of the presence or absence of diabetes mellitus or impaired glucose and will be evaluated twice: before and 6 months after efficient treatment of Cushing's syndrome. We make the hypothesis that Cushing's syndrome patients compared to healthy subjects have excess lipid storage in cardiac myocytes irrespectively of the glucose homeostasis status, and that this lipid content will decrease after the correction of hypercortisolism.

ELIGIBILITY:
Inclusion Criteria:

* group 1 and 2: patients with overt Cushing's syndrome, with 24-hour urinary free cortisol excretion over the two fold of the upper limit of the normal, with (group 1) or without (group 2) diabetes mellitus or glucose intolerance
* group 3: healthy volunteers matched for age, sex and BMI with the patients of the group 2

Exclusion Criteria:

* contraindication of MRI
* hypersensitivity to gadolinium
* acute myocardial ischemia
* renal insufficiency (creatinin clearance 30 mL/min/l,73m2)
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular (LV) intramyocardial triglyceride / water ratio LV intramyocardial triglyceride / water ratio | Assessed twice in patients - before and 6 months after treatment - and once in volunteers
  Intramyocardial triglyceride content will be assessed by 1H magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Left Ventricular intramyocardial fatt fraction (Dixon) | Assessed twice in patients - before and 6 months after treatment - and once in volunteers
  In/Out of Phase Imaging (Dixon)
Subcutaneous and visceral abdominal fatt | Assessed twice in patients - before and 6 months after treatment - and once in volunteers
  ISubcutaneous and visceral abdominal fat masses were determined from abdominal axial images at the L3 to L4 level
Cardiac morphology and function | Assessed twice in patients - before and 6 months after treatment - and once in volunteers
  LV mass index, LA, LV and Right Ventricular (RV) ejection fractions and LV and RV stroke volumes assessed by Cardiac Magnetic Resonance Imaging (CMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CHANSON, MD, PhD, Principal Investigator — AP-HP, Bicêtre Hospital
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Wolf P, Marty B, Bouazizi K, Kachenoura N, Piedvache C, Blanchard A, Salenave S, Prigent M, Jublanc C, Ajzenberg C, Droumaguet C, Young J, Lecoq AL, Kuhn E, Agostini H, Trabado S, Carlier PG, Feve B, Redheuil A, Chanson P, Kamenicky P. Epicardial and Pericardial Adiposity Without Myocardial Steatosis in Cushing Syndrome. J Clin Endocrinol Metab. 2021 Nov 19;106(12):3505-3514. doi: 10.1210/clinem/dgab556. PMID 34333603